CLINICAL TRIAL: NCT07200882
Title: Assessment of Tyrosine Kinase Inhibitors on Thyroid Functions in Patients With Chronic Myeloid Leukemia
Brief Title: What is the Impact of TKI on Thyroid Function in CML Patients?
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa salah sayed gaber, Resident in Hematology and Endocrinology units, Assiut University
Other Study IDs: TKI-CML
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Leukaemia (Chronic)
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the impact of various TKI on thyroid function in patients diagnosed with cml

DETAILED DESCRIPTION:
Tyrosine kinase inhibitors (TKIs) block the phosphorylation pathways of cellular signaling proteins, essential for tumor cell proliferation . Several endocrine side efects have been described with the increased use of TKIs in cancer therapy and thyroid alterations, mostly hypothyroidism, repre- sents a well-known phenomenon . TKI-induced thyroid alterations are caused by several direct mechanisms, such as thyroid damage ranging from mild follicular cells toxicity to destructive thyroiditis , inhibition of thyroid per- oxidase, blocking iodine uptake, and increased thyroid hor- mone clearance. TKIs may also induce indirect thy- roid damage via their antiangiogenic activity . More recently, de novo appearance of serum thyroid autoantibodies has been observed in almost one-third of oncologic patients followed before and during sunitinib therapy, suggesting that triggering of thyroid autoimmunity maybe involved in TKIs- induced thyroid dysfunction . Both hypothyroidism and thyroid autoimmunity induced by TKIs inpatients with diferent solid tumors have been found to be associated with a betteronc- ologic response, TKIs are routinely employed in the treatment of Philadel- phia chromosome-positive chronic myeloid leukemia (Ph- positive CML) . TheseTKIs specifcally target the oncogenic activity of the breakpoint cluster region (BCR)-Abelson murine leukemia viral oncogene homolog (ABL) protein in patients with CML. Four TKIs have been approved for frst- line therapy (FLT) CML: imatinib (frst-generation TKI), dasatinib, nilotinib, and bosutinib (second-generation TKI) . In cases of failure/resistance, all second-generation TKIs are efective, but the criteria for the choice of the second-line therapy (SLT) are patient related and depend on age, comor- bidities, and toxicity ofFLT with TKIs Besides a recent review of cases reported by the U.S. Food and Drug Admin- istration [20], only one retrospective monocentric study has been carried out on thyroid function in patients with CML on TKIs treatment [8], showing that thyroid dysfunction (mainly subclinical) is common during both frst-generation and second-generation TKIs therapy. However, no data are available on the relevance of thyroid autoimmunity in TKIs- induced thyroid dysfunction in patients with CML and on the potential relationship between thyroid dysfunction/auto- immunity and the response to treatment. With this concept in mind, we assessed thyroid function and autoimmunity in relation to the outcome of disease ina series of CML patients during treatment with frst- and second-generation TKIs.

ELIGIBILITY:
Inclusion Criteria:

* Patients age from 18 to 65 year

Newly diagnosed CML patients with Philadelphia chromosome positive based on peripheral blood findings and molecular analysis for the BCR-ABL mutation initiating ttt with a TKI (Philadelphia chromosome positive. CML patients )

Exclusion Criteria:

* -any history of using drugs interfering with TKI or having effect on thyroid function (Dexamethasone, Phenytoin, Carbamazepine, Rifampin and Phenobarbital)

Patients with a history of thyroid disease ( hypo or hyperthyroidism or auto immunity )or are already on treatment for thyroid dysfunction

* pregnancy and lactation
* concomitant use of oral contraceptive pills or corticosteroids.
* Other malignancies requiring concurrent treatment
* previous ttt with TKI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Philadelphia chromosome positive. CML patients
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
the impact of TKIs on thyroid in patients with Cml | 1 year
  To evaluate the impact of TKIs on thyroid in patients with Cml by measuring changes in thyroid
  hormone levels ( TSH
  Free T4
  Free T3)
  over time and determining the prevalence of thyroid disorder (hyperthyroidism and hypothyroidism )among tki treated patients